CLINICAL TRIAL: NCT02487225
Title: Pentoxifylline Treatment in Acute Pancreatitis: A Double-Blind Placebo - Controlled Randomized Trial
Brief Title: Pentoxifylline Treatment in Acute Pancreatitis (AP)
Acronym: AP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Santhi Swaroop Vege, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15-001710; 1R21DK101889-01A1 (NIH)
Record Dates: First submitted 2015-06-29; First posted 2015-07-01 (Estimated); Results first posted 2019-01-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Acute Pancreatitis (AP); Gallstone Pancreatitis; Alcoholic Pancreatitis; Trauma Acute Pancreatitis; Hypertriglyceridemia Acute Pancreatitis; Idiopathic (Unknown) Acute Pancreatitis; Medication Induced Acute Pancreatitis; Cancer Acute Pancreatitis; Miscellaneous (i.e. Acute on Chronic Pancreatitis)
Keywords: Post-Endoscopic Retrograde Cholangiopancreatography (ERCP) pancreatitis
MeSH Terms: conditions — Pancreatitis; Pancreatitis, Alcoholic | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pentoxifylline (Experimental): Pentoxifylline, 400 mg, 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects to receive up to a maximum of 9 doses.
  Interventions: Drug: Pentoxifylline
- Placebo (Placebo Comparator): Placebo 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects to receive up to a maximum of 9 doses.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pentoxifylline — Pentoxifylline is a competitive nonselective phosphodiesterase inhibitor which raises intracellular cyclic adenosine monophosphate (cAMP), activates protein kinase A (PKA), inhibits Tumor Necrosis Factor (TNF) and leukotriene synthesis, and reduces inflammation and innate immunity. In addition, pentoxifylline improves red blood cell deformability (known as a haemorrheologic effect), reduces blood viscosity and decreases the potential for platelet aggregation and thrombus formation.Pentoxifylline is also an antagonist at adenosine 2 receptors
  Other Names: Trental; Pentox; Pentoxil; Flexital
  Arms: Pentoxifylline
Drug: Placebo — A harmless pill that has no therapeutic effect, used as a control in testing of investigational drug
  Arms: Placebo

SUMMARY:
The purpose of this study was to determine the effects (good and bad) of giving a drug called pentoxifylline to patients with acute pancreatitis.

DETAILED DESCRIPTION:
Participants were randomized to either the treatment group (Pentoxifylline medication) or the control group (Placebo).

Participant took a pill orally, starting from the time of admission. Participants received a total of 9 doses over the three days of hospitalization (72 hours).

Research blood draws were done at baseline and on 5 successive days or until the time of discharge, whichever occured earlier. The study gathered clinical follow up information up to 4 months following hospitalization regarding the diagnosis of acute pancreatitis.

ELIGIBILITY:
Inclusion criteria

* Enrollment within 72 hours of diagnosis of acute pancreatitis (AP)
* Ability to give informed consent or a Legal Adult Representative (LAR) able to give informed consent for subject when needed as defined buy LAR use guidelines.
* Adult subjects of age ≥18 years.

Exclusion Criteria:

* Moderate or severe congestive heart failure
* History of seizure disorders or demyelinating disease
* Nursing mothers
* Pregnancy
* History of prior tuberculosis or risk factors for tuberculosis
* Evidence of non- corticosteroid immunosuppression (such as malignancy, chronic renal failure, chemotherapy within 60 days, and HIV)
* Evidence of active hemorrhage
* Paralytic ileus with severe nausea and vomiting

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2015-05; Primary Completion 2017-04-30 (Actual); Study Completion 2017-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Santhi Swaroop Vege, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at Mayo Clinic in Rochester, Minnesota.
Groups:
- Pentoxifylline: Pentoxifylline, 400 mg, 3 times daily by mouth from time of enrollment until 72 hours from enrollment. Subjects to receive up to a maximum of 9 doses.
  Pentoxifylline: Pentoxifylline is a competitive nonselective phosphodiesterase inhibitor which raises intracellular cyclic adenosine monophosphate (cAMP), activates protein kinase A (PKA), inhibits TNF and leukotriene synthesis, and reduces inflammation and innate immunity. In addition, pentoxifylline improves red blood cell deformability (known as a haemorrheologic effect), reduces blood viscosity and decreases the potential for platelet aggregation and thrombus formation.Pentoxifylline is also an antagonist at adenosine 2 receptors
Period: Overall Study
Arm/Group | Pentoxifylline | Placebo
Started | 45 | 38
Completed | 18 | 8
Not Completed | 27 | 30

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pentoxifylline | Placebo | Total
Number analyzed (Participants) | 45 | 38 | 83
Age, Continuous [Median (Full Range); unit: years] | 63.0 [23.0 to 86.0] | 55.5 [23.0 to 81.0] | 59.0 [23.0 to 86.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 24 | 17 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 2 | 0 | 2
  White | 41 | 36 | 77
  Other | 2 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 45 | 38 | 83
Bedside Index of Severity in Acute Pancreatitis (BISAP) Score [Median (Full Range); unit: units on a scale] — A scale of 0-5 used to predict mortality in patients with acute pancreatitis. A score of 0-2 is low mortality of less than 2%. A score of 3-5 is associated with higher mortality of more than 15%.
  units on a scale | 1.0 [0.0 to 2.0] | 0.5 [0.0 to 2.0] | 1.0 [0.0 to 2.0]
Systematic Inflammatory Response Syndrome (SIRS) score on admission [Median (Full Range); unit: units on a scale] — Sepsis is an infection which as evoked a systemic inflammatory response. Clinically, the Systemic Inflammatory Response Syndrome (SIRS) is identified by two or more symptoms including fever or hypothermia, tachycardia, tachypnea and change in blood leucocyte count. Measurements are made on a scale from 0 to 4, with higher scores indicating more severe failure symptoms.
  units on a scale | 1.0 [0.0 to 3.0] | 1.0 [0.0 to 4.0] | 1.0 [0.0 to 4.0]

OUTCOME MEASURES:

1. Primary Outcome: Change in C-reactive Protein (C-RP) From Admission Baseline at One Week.
Description: C-reactive protein is a substance produced by the liver in response to inflammation. Normal C-RP levels are below 3.0 mg/L.Units: mg/L
Time Frame: Admission (baseline), day 5
Population: Eighteen (18) of forty-five subjects (45) in the treatment arm and eight (8) of thirty-eight (38) subjects in the placebo arm completed the study. Additionally, subjects had blood collections for 5 days or until dismissal. Many subjects were dismissed at 2-3 days.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 45 | 38
mg/L
  Admission (baseline) | 86.2 (81.5) | 75.8 (83.1)
  Day 5: number analyzed (Participants) | 9 | 5
  Day 5 | 116.4 (100.4) | 127.2 (97.8)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Admission (baseline); Test type: Superiority; p = 0.5796, Kruskal-Wallis
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Day 5; Test type: Superiority; p = 0.8415, Kruskal-Wallis

2. Primary Outcome: Change in Tumor Necrosis Factor-alpha (TNF-a) Levels From Admission Baseline at One Week.
Description: Tumor Necrosis Factor Alpha is a cell signaling protein (cytokine) involved in systemic inflammation and is one of the cytokines that make up the acute phase reaction. TNF is important to the body because it helps regulate the response of the immune system to a foreign object, especially to the present cancerous tumor. It promotes inflammation, produces other cells used in the inflammatory response, and can help cells heal. The normal range is 5 to 27.2 pg/ml.Units: pg/ml
Time Frame: Admission (baseline), day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 40 | 37
pg/ml
  Admission (baseline) | 1.9 (0.9) | 1.8 (1.3)
  Day 5: number analyzed (Participants) | 9 | 5
  Day 5 | 4.3 (6.3) | 1.9 (0.7)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Admission (baseline); Test type: Superiority; p = 0.1109, Kruskal-Wallis
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Test type: Superiority; p = 0.4619, Kruskal-Wallis

3. Primary Outcome: Change in Interleukin-6 (IL-6) Levels From Admission Baseline at One Week.
Description: Interleukin-6 (IL-6) may be used to help evaluate a person who has a condition associated with inflammation, such as lupus or rheumatoid arthritis, or with infection, such as sepsis. It may also be used in the evaluation of diabetes or cardiovascular disease. IL-6 is a cytokine, a protein produced by immune cells that acts on other cells to help regulate and/or promote an immune response. It also stimulates the production of acute phase reactants, proteins that increase in the blood with conditions that cause inflammation or tissue injury. Circulating IL-6 can be found in the blood of normal individuals in the 1 pg/mL range, with slight elevations during the menstrual cycle, modest elevations in certain cancers (melanoma) (10 pg/mL), and large elevations after surgery (30-430 pg/mL).Units: pg/ml
Time Frame: Admission (baseline), day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 42 | 35
pg/mL
  Admission (baseline) | 107.9 (124.8) | 89.1 (138.2)
  Day 5: number analyzed (Participants) | 9 | 5
  Day 5 | 81.8 (97.4) | 88.6 (85.2)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Admission (baseline); Test type: Superiority; p = 0.1236, Kruskal-Wallis
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Day 5; Test type: Superiority; p = 0.9468, Kruskal-Wallis

4. Primary Outcome: Change in Interleukin-8 (IL-8) Levels From Admission Baseline at One Week.
Description: IL-8 is a chemotactic factor that attracts neutrophils, basophils, and T-cells, but not monocytes. It is also involved in neutrophil activation. It is released from several cell types in response to an inflammatory stimulus. Units: pg/mL
Time Frame: Admission (baseline), day 5
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Pentoxifylline | Placebo
Number analyzed (Participants) | 42 | 36
pg/ml
  Admission (baseline) | 43.7 (29.4) | 31.5 (26.1)
  Day 5: number analyzed (Participants) | 9 | 5
  Day 5 | 45.9 (43.2) | 32.1 (23.5)
Statistical Analysis 1: Comparison: Pentoxifylline vs Placebo; Admission (baseline); Test type: Superiority; p = 0.157, Kruskal-Wallis
Statistical Analysis 2: Comparison: Pentoxifylline vs Placebo; Day 5; Test type: Superiority; p = 0.3173, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: 4 months
Arm/Group | Pentoxifylline | Placebo
All-Cause Mortality (participants affected / at risk) | 2/45 | 0/38
Serious Adverse Events (participants affected / at risk) | 1/45 | 0/38
Other Adverse Events (participants affected / at risk) | 12/45 | 5/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline (N=45) | Placebo (N=38)
Hospitalized for psychological evaluation, considered a danger to self (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pentoxifylline (N=45) | Placebo (N=38)
Sepsis due to disease progression (General disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Headache/Migraine (General disorders) | 1 (1) | 2 (2)
Angina (Cardiac disorders) | 2 (2) | 0
Necrosis due to disease progression (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Infected cystic duct leak (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hip pain and gait dysfunction (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-09): https://cdn.clinicaltrials.gov/large-docs/25/NCT02487225/Prot_SAP_000.pdf